CLINICAL TRIAL: NCT07015710
Title: Impact of Gamma Knife Radiosurgery on Tectal Plate Gliomas
Brief Title: Gamma Knife Radiosurgery on Tectal Plate Gliomas
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Awad Mohamed Hegab, Lecturer of Neurosurgery, Faculty of Medicine, Al-Azhar University, Damietta, Egypt., Al-Azhar University
Other Study IDs: DFM-IRB 00012367-25-05-007
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Gamma Knife Radiosurgery; Tectal Plate Gliomas
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tectal Plate Gliomas group: Patients underwent gamma knife radiosurgery (GKRS) for tectal plate gliomas (TPGs).
  Interventions: Procedure: Gamma Knife Radiosurgery

INTERVENTIONS:
Procedure: Gamma Knife Radiosurgery — Patients underwent gamma knife radiosurgery (GKRS) for tectal plate gliomas (TPGs).

SUMMARY:
This study aimed to assess the impact of gamma knife radiosurgery on tectal plate gliomas (TPGs).

DETAILED DESCRIPTION:
Tectal plate gliomas (TPGs) represent a subset of brainstem gliomas that are predominantly slow-growing, low-grade tumors and rarely produce neurological deficits.

Viable options include biopsy and monitoring with serial neuroimaging, surgical resection, radiotherapy (either early following surgery or late on evidence of disease progression), chemotherapy, and stereotactic radiosurgery (SRS).

SRS using Gamma Knife radiosurgery (GKRS) has been identified in small case series as a safe and promising approach for managing TPGs that necessitate intervention beyond mere observation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 5 to 55 years.
* Both sexes.
* Patients underwent gamma knife radiosurgery (GKRS) for tectal plate gliomas (TPGs).

Exclusion Criteria:

* High-grade glioma.
* Tumor extension beyond the tectal region.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This retrospective study will be conducted in the Department of Neurosurgery, Al-Azhar University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of response | One year post-procedure
  Incidence of response was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University (Damietta), Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.